CLINICAL TRIAL: NCT02712372
Title: A Phase I, Randomised, Single-Blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD4831 After Single and Multiple Ascending Dose Administration to Healthy Male Subjects
Brief Title: A Study to Assess the Safety and Tolerability of Single and Multiple Doses of AZD4831 in Healthy Male Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D6580C00001
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Cardiovascular Disease
Keywords: AZD4831 oral suspension; Healthy male subjects; Safety; Tolerability; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Cardiovascular Diseases | interventions — AZD4831

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (10):
- Part 1, Dose Level 1 (Experimental): Part 1: Part 1A: Single dose administered in the morning on Day 1 under fasted conditions. Part 1B: Single dose administered in the morning of Day 1 under fed conditions.
  Interventions: Drug: AZD4831
- Part 1, Dose Level 2 (Experimental): Part 1: Part 1A: Single dose administered in the morning on Day 1 under fasted conditions. Part 1B: Single dose administered in the morning of Day 1 under fed conditions.
  Interventions: Drug: AZD4831
- Part 1, Dose Level 3 (Experimental): Part 1: Part 1A: Single dose administered in the morning on Day 1 under fasted conditions. Part 1B: Single dose administered in the morning of Day 1 under fed conditions.
  Interventions: Drug: AZD4831
- Part 1, Dose Level 4 (Experimental): Part 1: Part 1A: Single dose administered in the morning on Day 1 under fasted conditions. Part 1B: Single dose administered in the morning of Day 1 under fed conditions.
  Interventions: Drug: AZD4831
- Part 1, Dose Level 5 (Experimental): Part 1: Part 1A: Single dose administered in the morning on Day 1 under fasted conditions. Part 1B: Single dose administered in the morning of Day 1 under fed conditions.
  Interventions: Drug: AZD4831
- Part 1, Dose Level 6 (Experimental): Part 1: Part 1A: Single dose administered in the morning on Day 1 under fasted conditions. Part 1B: Single dose administered in the morning of Day 1 under fed conditions.
  Interventions: Drug: AZD4831
- Part 2, Dose Level 1 (Experimental): Part 2: Single dose administered in the morning on Day 1 and multiple doses administered once daily, in the morning, Days 3 to 12
  Interventions: Drug: AZD4831
- Part 2, Dose Level 2 (Experimental): Part 2: Single dose administered in the morning on Day 1 and multiple doses administered once daily, in the morning, Days 3 to 12
  Interventions: Drug: AZD4831
- Part 2, Dose Level 3 (Experimental): Part 2: Single dose administered in the morning on Day 1 and multiple doses administered once daily, in the morning, Days 3 to 12
  Interventions: Drug: AZD4831
- AZD4831 Placebo (Placebo Comparator): Part 1: Part 1A: Single dose administered in the morning on Day 1 under fasted conditions. Part 1B: Single dose administered in the morning of Day 1 under fed conditions.
  Part 2: Single dose administered in the morning on Day 1 and multiple doses administered once daily, in the morning, Days 3 to 12
  Interventions: Drug: AZD4831 placebo

INTERVENTIONS:
Drug: AZD4831 — AZD4831 1-50 mg/g oral suspension
  Arms: Part 1, Dose Level 1; Part 1, Dose Level 2; Part 1, Dose Level 3; Part 1, Dose Level 4; Part 1, Dose Level 5; Part 1, Dose Level 6; Part 2, Dose Level 1; Part 2, Dose Level 2; Part 2, Dose Level 3
Drug: AZD4831 placebo — AZD4831 placebo oral suspension
  Arms: AZD4831 Placebo

SUMMARY:
This is a Phase I, first-in-human (FIH) study to assess the safety, tolerability, pharmacokinetics (PK) and Pharmacodynamics (PD) of AZD4831 after single and multiple ascending doses in healthy male subjects

DETAILED DESCRIPTION:
This is a Phase I, FIH, randomized, single-blind, placebo-controlled study to assess the safety, tolerability, pharmacokinetics (PK) and Pharmacodynamics (PD) of AZD4831 after single (Part 1) and multiple (Part 2) ascending doses in healthy male subjects. The study will be conducted at a single study center with a planned number of subjects of up to 125 healthy males, aged 18 to 50 years.

ELIGIBILITY:
Inclusion Criteria

* Provision of signed and dated, written informed consent before any study specific procedures.
* Healthy male subjects aged 18 - 50 years, inclusive, with suitable veins for cannulation or repeated venipuncture.
* Have a body mass index (BMI) between 18 and 29.9 kg/m2, inclusive, and weigh at least 50 kg and no more than 100 kg inclusive.
* Provision of signed, written and dated informed consent for optional genetic/biomarker research.
* Subjects must be able to read, speak and understand the German language.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Presence of infection(s) (particularly fungal infection), as judged by the investigator.
* History or current thyroid disease.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational medicinal product (IMP).
* Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, as judged by the investigator.
* Any positive result on screening for serum hepatitis B surface antigen (HBsAg), anti-hepatitis B core (anti-HBc) antibodies, hepatitis C antibody and human immunodeficiency virus (HIV).
* Abnormal vital signs
* Any clinically significant abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically significant abnormalities in the 12-lead ECG, as considered by the investigator that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or LV hypertrophy.
* Prolonged QTcF > 450 ms or shortened QTcF < 340 ms or family history of long QT syndrome.
* PR(PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation)
* PR (PQ) interval prolongation (> 200 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third degree AV block, or AV dissociation
* Persistent or intermittent complete bundle branch block, incomplete bundle branch block, or intraventricular conduction delay with QRS > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of, for example, ventricular hypertrophy or pre-excitation.
* ECG findings suggesting a metabolic or other non-cardiac condition that may confound interpretation of serial changes (such as hypokalemia).
* Known or suspected history of drug abuse, as judged by the investigator.
* Current smokers or those who have smoked or used nicotine products within the previous 3 months.
* History of alcohol abuse or excessive intake of alcohol, as judged by the investigator.
* Positive screen for drugs of abuse, cotinine (nicotine) or alcohol at screening or admission to the unit before the first administration of IMP.
* History of severe allergy/hypersensitivity or ongoing clinically significant allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD4831.
* Excessive intake of caffeine containing drinks or food (e.g., coffee, tea, chocolate), as judged by the investigator.
* Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks before the first administration of IMP.
* Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks before the first administration of IMP or longer if the medication has a long half-life.
* Plasma donation within 1 month of screening or any blood donation/blood loss > 500 mL during the 3 months before screening.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest.
* Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
* Involvement of any Astra Zeneca, PAREXEL or study site employee or their close relatives.
* Judgment by the investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
* Subjects who are vegans or have medical dietary restrictions.
* Subjects who cannot communicate reliably with the investigator.

Exclusion from the genetic research:

* Previous bone marrow transplant.
* Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2016-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Frequencies of adverse events | From screening up to 10 days post final dose
  To assess the safety and tolerability of single and multiple doses of AZD4831
Supine blood pressure (Part 1) | From screening up to 48 hours post dose
  To assess change from baseline in supine blood pressure
Supine pulse rate (Part 1) | From screening up to 48 hours post dose
  To assess change from baseline in supine pulse rate
Supine body temperature (Part 2) | From screening up to pre-dose Day 12
  To assess change from baseline in supine body temperature
12-lead electrocardiogram | From screening up to 10 days post final dose
  To assess 12-lead electrocardiogram
12-lead electrocardiogram (cardiac telemetry) | From Day-1 up to 24 hours post final dose
  12-lead electrocardiogram (cardiac telemetry)
Physical examination | From screening up to 10 days post final dose
  To assess subject through a physical examination, including assessment of the general appearance, skin, cardiovascular, respiratory, abdomen, head and neck (including ears, eyes, nose and throat), lymph nodes, thyroid, musculoskeletal and neurological systems.
To assess the subject through hematology laboratory assessment | From screening up to 10 days post final dose
  To assess a subject through hematology laboratory assessment
Percentage of adverse events | From screening to 10 days post final dose
  To assess the safety and tolerability of single and multiple doses of AZD4831
Supine blood pressure (Part 2) | From screening up to 10 days post final dose
  To assess change from baseline in supine blood pressure
Supine pulse rate (Part 2) | From screening up to 10 days post final dose
  To assess change from baseline in supine pulse rate
Chemistry evaluations | From screening up to 10 days post final dose
  including high-sensitivity C-reactive protein {hs-CRP} and thyroid panel
To assess the subject through urinalysis laboratory assessment | From screening up to 10 days post final dose
  To assess a subject through urinalysis laboratory assessment

SECONDARY OUTCOMES:
Observed maximum plasma concentration, taken directly from the individual concentration-time curve (Cmax) | From pre-dose up to 48 hours post dose
  To characterize the plasma pharmacokinetics of AZD4831
Time to reach maximum plasma concentration, taken directly from the individual concentration-time curve (tmax) | From pre-dose up to 48 hours post dose
  To characterize the plasma pharmacokinetics of AZD4831
Terminal rate constant, estimated by log-linear least squares regression of the terminal part of the concentration-time curve (λz) | From pre-dose up to 48 hours post dose
  To characterize the plasma pharmacokinetics of AZD4831
Terminal half-life, estimated as (ln2)/λz (t1/2λz) | From pre-dose up to 48 hours post dose
  To characterize the plasma pharmacokinetics of AZD4831
Area under the plasma concentration-curve over 24 hours (AUCτ) | From pre-dose up to 48 hours post dose
  To characterize the plasma pharmacokinetics of AZD4831
Area under the plasma concentration-curve from time zero to the time of last quantifiable analyte concentration (AUC0-t) | From pre-dose up to 48 hours post dose
  To characterize the plasma pharmacokinetics of AZD4831
Area under the concentration-time curve from time zero extrapolated to infinity (AUC) | From pre-dose up to 48 hours post dose
  To characterize the plasma pharmacokinetics of AZD4831
Apparent clearance for parent drug estimated as dose divided by AUC (CL/F) | From pre-dose up to 48 hours post dose
  To characterize the plasma pharmacokinetics of AZD4831
Mean Residence Time (MRT) | From pre-dose up to 48 hours post dose
  To characterize the plasma pharmacokinetics of AZD4831
Apparent volume of distribution for parent drug at terminal phase (Vz/F) | From pre-dose up to 48 hours post dose
  To characterize the plasma pharmacokinetics of AZD4831
Area under the plasma concentration-time curve from time zero to time of last quantifiable analyte concentration divided by the dose administered (AUC0-t/D) | From pre-dose up to 48 hours post dose
  To characterize the plasma pharmacokinetics of AZD4831
Area under the plasma concentration-time curve from time zero extrapolated to infinity divided by the dose administered (AUC/D) | From pre-dose up to 48 hours post dose
  To characterize the plasma pharmacokinetics of AZD4831
Observed maximum plasma concentration divided by the dose administered (Cmax/D) | From pre-dose up to 48 hours post dose
  To characterize the plasma pharmacokinetics of AZD4831
Area under the plasma concentration-curve over the dosing interval divided by the dose administered (AUCτ/D) (Part 2 only) | From pre-dose up to 48 hours post final dose
  To characterize the plasma pharmacokinetics of AZD4831
Accumulation ratio calculated as AUCτ Day 12/ AUCτ Day 1 (Rac AUC) (Part 2 only) | From pre-dose up to 48 hours post final dose
  To characterize the plasma pharmacokinetics of AZD4831
Accumulation ratio calculated as Cmax Day 12/ Cmax Day 1 (Rac Cmax) (Part 2 only) | From pre-dose up to 48 hours post final dose
  To characterize the plasma pharmacokinetics of AZD4831
Temporal change parameter in systemic exposure (TCP) (Part 2 only) | From pre-dose up to 48 hours post final dose
  To characterize the plasma pharmacokinetics of AZD4831
Amount of analyte excreted into the urine from time t1 to t2 [Ae(t1-t2)] | From pre-dose up to 48 hours post dose
  Assessment of the urine PK following single and multiple doses of pharmacokinetics of AZD4831
Cumulative amount of analyte excreted at time t [Ae(0-t)] | From pre-dose up to 48 hours post dose
  Assessment of the urine PK following single and multiple doses of pharmacokinetics of AZD4831
Fraction of dose excreted unchanged into the urine from time t1 to t2, estimated by dividing Ae(t1-t2) by dose [fe(t1-t2)] | From pre-dose up to 48 hours post dose
  Assessment of the urine PK following single and multiple doses of pharmacokinetics of AZD4831
Fraction of dose excreted unchanged into the urine from time zero to time t, estimated by dividing Ae(0-t) by dose [fe(0-t)] | From pre-dose up to 48 hours post dose
  Assessment of the urine PK following single and multiple doses of pharmacokinetics of AZD4831
Renal clearance, estimated by dividing Ae(0-t) by AUC(0-t) (CLR) | From pre-dose up to 48 hours post dose
  Assessment of the urine PK following single and multiple doses of pharmacokinetics of AZD4831

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, Dr. med., Principal Investigator — PAREXEL Early Phase Clinical Unit Berlin, On the premises of Klinikum Westend, Haus 31, Spandauer Damm 130, 14050 Berlin, Germany